CLINICAL TRIAL: NCT03872765
Title: Cohort Study of Chronic Anal Fissure Management Using CO2 Laser
Brief Title: Outcomes of the Use of CO2 (Carbon Dioxide) Laser in the Treatment of Chronic Anal Fissure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nineveh (Other)
Responsible Party: Principal Investigator, Ahmed Haidaran, Consultant general surgeon, lecturer, University of Nineveh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 818965
Record Dates: First submitted 2019-01-13; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Chronic Anal Fissure
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with chronic anal fissure (Other): Use of laser in surgery of chronic anal fissure instead of the conventional surgical techniques.
  Interventions: Device: Laser surgery

INTERVENTIONS:
Device: Laser surgery — Use of CO2 laser to perform surgeries to treat chronic anal fissure

SUMMARY:
Outcomes of using CO2 (Carbon Dioxide) laser in the management of chronic anal fissure as an alternative to conventional methods

DETAILED DESCRIPTION:
The use of CO2 laser in management of chronic anal fissure as a new alternative technique. Interventional study of 236 patients. Comparison to other techniques was made with respect to pain scores and healing time.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic anal fissure

Exclusion Criteria:

* Acute anal fissure Pregnancy

Ages: 26 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 236 (Actual)
Dates: Start 2012-01-14 (Actual); Primary Completion 2014-09-09 (Actual); Study Completion 2014-09-09 (Actual)

PRIMARY OUTCOMES:
Pain score after surgery (Degree of pain) | 3 weeks after surgery
  Record pain after surgery on a scale of 1 to 10 (Range 1-10 with 1 being least pain and 10 greatest pain experienced by patients)
Recovery time after surgery (How many days patient takes to recover) | 3 weeks
  Time (How many days) for patient to be able to return to normal life activities after surgery
Incontinence after surgery | 2 years
  Lack of control of anal sphincter (Incontinence)

IPD SHARING:
Plan to Share IPD: No